CLINICAL TRIAL: NCT07323186
Title: Evaluation of the NEOmom® Gastric Video Capsule for Gastric Cancer Screening
Acronym: NEOTOGAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC25_0258
Record Dates: First submitted 2025-12-04; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Stomach Cancer; Diagnosis; Endoscopy of Stomach (Procedure)
Keywords: stomach cancer
MeSH Terms: conditions — Stomach Neoplasms; Disease | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- magnetically controlled video capsule endoscope + Standard EGD (Experimental): Participants undergo both magnetically controlled video capsule endoscopy and standard oesophagogastroduodenal endoscopy during the same visit, allowing intra-patient comparison of lesion detection.
  Interventions: Device: Magnetically controlled video capsule endoscopy (MC-VCE)

INTERVENTIONS:
Device: Magnetically controlled video capsule endoscopy (MC-VCE) — -Intervention 1 description: Ingestion of the NEOMOM® magnetically controlled video capsule, guided by an external magnetic field and coupled with an artificial intelligence module to ensure completeness of gastric examination and assist in lesion detection.
  -Intervention 2 Description: Conventional oesophagogastroduodenal endoscopy performed according to standard clinical practice.

SUMMARY:
Gastric cancer remains a major public health concern, with approximately 6,600 new cases diagnosed each year in France. Despite therapeutic progress, its overall prognosis is still poor: the 5-year survival rate across all stages remains below 30%. This survival is closely linked to the stage at diagnosis. Early-stage gastric cancer has an excellent prognosis, with survival rates above 90%, while advanced-stage disease shows survival below 10%. This dramatic contrast underscores the critical need to develop and implement approaches that enable earlier and more reliable diagnosis. Early detection is therefore one of the most powerful strategies to reduce mortality from this severe and often silent disease.

Within this context, the overall ambition of the NEOTOGAS project is to contribute to lowering gastric-cancer mortality by improving the ability to diagnose the disease at an early, more treatable stage. The project positions itself within the broader field of prevention, targeting one of the leading and most challenging public health issues. Gastric cancer is often a potentially fatal condition that typically develops over many years, most commonly as a consequence of chronic infection with Helicobacter pylori (H. pylori). Identifying precancerous gastric lesions before the appearance of invasive cancer thus represents a strategic priority for the healthcare system.

Our central hypothesis is that a non-invasive, robot-assisted endoscopic approach using a magnetic-guided capsule-the NEOMOM system-will prove effective for detecting precancerous gastric lesions. If validated, this technology could form the foundation of an organized, large-scale screening program. Such a screening strategy would represent a major innovation, particularly in populations at higher risk due to H. pylori infection or other predispositions. The ability to offer a less invasive, more accessible examination could significantly increase screening adherence and facilitate earlier diagnosis.

The NEOTOGAS study is based on an innovative combination of technologies: a magnetic-guided videocapsule steered inside the stomach using the NEOMOM robot, supported by artificial intelligence to assist image acquisition and interpretation. The study aims to assess the level of concordance between lesion detection through the current gold-standard procedure (conventional endoscopy) and this new capsule-based examination. Beyond diagnostic performance, the project also integrates several essential dimensions for future implementation: patient acceptability of the procedure, overall cost, duration of the examination, and the potential clinical and organizational benefits of this alternative approach.

A key component of the project is the creation of high-quality image banks. These will support the development of advanced AI models capable of enhancing lesion detection and ensuring the completeness of the stomach examination. Such resources will be instrumental in evaluating whether magnetic-guided capsule endoscopy could realistically be integrated into structured gastric cancer screening pathways in the future. The project therefore aims not only to evaluate a device, but also to explore its broader screening potential and its capacity to transform clinical practice.

The primary objective of the NEOTOGAS study is to rigorously assess the performance of this innovative medical device, which combines magnetic navigation with AI-assisted image interpretation, in detecting gastric lesions. The AI module plays a dual role: ensuring that the entire stomach is adequately explored and helping highlight images of interest for clinicians during analysis. By improving both completeness and accuracy, the technology could represent a significant advancement over existing non-invasive diagnostic tools.

To achieve these goals, the study plans to include a total of 100 patients over a 6-month period. This sample size will allow a robust comparison of diagnostic concordance while providing sufficient data to evaluate feasibility, patient experience, and operational parameters. The findings of NEOTOGAS will determine whether magnetic-guided capsule endoscopy can be considered a relevant and effective method for future organized gastric cancer screening programs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient,
* Aged between 50 and 74 inclusive with a life expectancy of at least 10 years,
* Undergoing screening or surveillance colonoscopy (for colorectal cancer or polyps)
* Patient who has received verbal and written information as well as a patient booklet on the VCE-CM examination and has given their written informed consent.
* Patient affiliated with a social security scheme
* Effective contraception throughout the study for women of childbearing age

Exclusion Criteria:

* Patients who have had or currently have the following (items from the TOGAS pilot study/specific to endoscope use) will not be included in the study:
* An EOGD in a high-volume endoscopy centre within the last 3 years
* Known gastric cancer
* Known genetic cancer syndromes
* Previous gastrectomy or bariatric gastric surgery
* Known gastric precancerous condition (gastric atrophy, intestinal metaplasia, dysplasia)
* Acute gastrointestinal haemorrhage in the last 4 weeks
* A coagulation disorder or medication that prevents biopsy sampling
* A risk associated with sedation or anaesthesia
* Severe heart disease
* An inability to actively consent to participation in the study, and patients under guardianship or legal protection.

Pregnant or breastfeeding patients will not be included.

Patients with the following conditions (specific to VCE-CM examination) will not be included in the study:

* Swallowing disorders or known gastroparesis
* A history of digestive surgery
* Clinical or radiological signs suggestive of narrowing of the digestive tract
* An occlusive or sub-occlusive condition, a known or suspected history of stenosis or digestive fistula
* Left heart failure with orthopnoea
* Overweight (> 135 kg)
* Reduced mobility (i.e. unable to transfer or move themselves)
* Persons with pacemakers, defibrillators or metallic foreign bodies (with the exception of dental implants) will not be included in order to avoid interference with the robot.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-07 (Estimated)

PRIMARY OUTCOMES:
Lesion-level concordance in gastric lesion detection between magnetic-controlled video capsule endoscopy and standard oesophagogastroduodenal endoscopy | Periprocedural (during the study visit) through image review within 72 hours after the examination (up to Day 8 in case of delayed capsule excretion)
  Lesion-level concordance between magnetic-controlled video capsule endoscopy (MC-VCE) and standard oesophagogastroduodenal endoscopy (EGD) for the detection of gastric lesions.
  Concordance will be expressed as agreement between the two modalities based on paired lesion detection (presence/absence), using expert review of recorded examinations.
  In case of discordant findings, an independent adjudication committee composed of two expert clinicians blinded to the initial readings will determine the final classification.

SECONDARY OUTCOMES:
Completeness of gastric examination assessed by magnetic-controlled video capsule endoscopy compared with standard oesophagogastroduodenal endoscopy | Periprocedural (during the study visit) through image review within 72 hours after the examination
  Proportion of complete gastric examinations achieved with magnetic-controlled video capsule endoscopy, as assessed by expert clinicians and compared with standard oesophagogastroduodenal endoscopy.
  Completeness is defined as visualization of all predefined gastric anatomical regions.
Lesion-by-lesion diagnostic performance of magnetic-controlled video capsule endoscopy compared with standard oesophagogastroduodenal endoscopy | Periprocedural (during the study visit) through image review within 72 hours after the examination
  Lesion-by-lesion diagnostic performance of magnetic-controlled video capsule endoscopy compared with standard oesophagogastroduodenal endoscopy, expressed as sensitivity, specificity, positive predictive value, and negative predictive value, using EGD as the reference standard.
Diagnostic performance of magnetic-controlled video capsule endoscopy for major gastric lesions compared with standard oesophagogastroduodenal endoscopy | Periprocedural (during the study visit) through image review within 72 hours after the examination
  Diagnostic performance of magnetic-controlled video capsule endoscopy for predefined major gastric lesions (gastric tumors, gastric ulcers, gastric cancer), expressed as sensitivity, specificity, positive predictive value, and negative predictive value, using standard oesophagogastroduodenal endoscopy as the reference standard.
Concordance between expert reading and artificial intelligence-assisted reading of magnetic-controlled video capsule endoscopy images | Image review within 72 hours after the examination
  Lesion detection concordance between conventional expert clinician reading and automated reading using the artificial intelligence module (Vue Smart V7 software) applied to magnetic-controlled video capsule endoscopy images.
  Diagnostic performance will be expressed as sensitivity, specificity, positive predictive value, and negative predictive value of AI-assisted reading compared with expert clinician interpretation
Diagnostic concordance between non-invasive blood tests combined with magnetic-controlled video capsule endoscopy and biopsies combined with standard oesophagogastroduodenal endoscopy | Periprocedural (during the study visit) through availability of histological results (up to Day 8)
  Diagnostic concordance between magnetic-controlled video capsule endoscopy combined with predefined non-invasive blood tests and standard oesophagogastroduodenal endoscopy combined with gastric biopsies, based on final diagnostic classification
Patient-reported acceptability score of magnetic-controlled video capsule endoscopy | Within 24 hours after completion of the magnetic-controlled video capsule endoscopy
  Patient-reported acceptability of magnetic-controlled video capsule endoscopy measured using a structured questionnaire with an ordinal scale.
  Scores range from 0 to 10, with higher scores indicating better acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No